CLINICAL TRIAL: NCT01484691
Title: Role of miRNAs in Th2-driven Inflammation in Asthma
Brief Title: Role of microRNAs in T Cell-Driven Inflammation in Asthma
Acronym: RITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-07039
Record Dates: First submitted 2011-10-26; First posted 2011-12-02 (Estimated); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy non-asthmatic controls (No Intervention): Healthy non-asthmatic controls who will be studied at one point in time and serve as a control group for the baseline bronchoscopy and evaluation of T-cell miRNA expression.
- Asthmatics (treatment) (Active Comparator): Steroid-naïve asthma (randomized to 8 weeks of treatment with inhaled corticosteroids). Asthmatics not on inhaled corticosteroids, randomized to inhaled budesonide, 1 puff (180mcg) twice a day for 8-10 weeks. These subjects will undergo bronchoscopy and T-cell miRNA measurement at baseline (before corticosteroids) and again after treatment with inhaled corticosteroids.
  Interventions: Drug: Budesonide
- Asthmatics (no treatment) (No Intervention): Steroid-naïve asthma (randomized to 8 weeks of no inhaled corticosteroid treatment). Asthmatics not on inhaled corticosteroids, randomized to no change in treatment for 8-10 weeks. These subjects will undergo bronchoscopy and T-cell miRNA measurement at baseline and again after 8 weeks without treatment with inhaled corticosteroids.

INTERVENTIONS:
Drug: Budesonide — Inhaled powder of inhaled corticosteroid, 1 puff (180mcg) twice a day for 8-10 weeks
  Other Names: Pulmicort
  Arms: Asthmatics (treatment)

SUMMARY:
This will be a single center study of asthmatic subjects and healthy controls which will investigate mechanisms of asthma through detailed molecular analysis of airway tissues and fluids. The primary goal will be investigate the role of microRNAs in Th2-driven inflammation in asthma. The investigators hypothesize that asthma is associated with abnormal expression of miRNAs in T cells which favors differentiation into Th2-cells. The investigators further hypothesize that asthma is heterogeneous based on the presence and absence of Th2-driven inflammation and that abnormalities in T cell miRNA expression will be most prominent in a subgroup with high levels of Th2-driven inflammation (as assessed using molecular markers that the investigators have previously established). Finally, the investigators hypothesize that inhaled corticosteroids will normalize the T-cell miRNA abnormalities observed in asthma, as corticosteroids treat Th2-driven inflammation. The samples collected will also facilitate the pursuit of secondary analyses designed to investigate mechanisms of inflammation and remodeling in asthma as well as molecular phenotypes of asthma.

ELIGIBILITY:
Group A:

Inclusion Criteria:

* Male and female subjects between the ages of 18 and 70 years

Group B:

Inclusion Criteria:

* Male and female subjects between the ages of 18 and 70 years
* History of asthma
* No use of oral or inhaled corticosteroids for the treatment of asthma in the past 6 weeks
* Hyperreactivity to methacholine (PC20FEV1 Methacholine ≤ 8.0 mg/mL)
* At least one of the following symptoms, beta agonist use, or FEV1 criteria:

  * Asthma symptoms on at least two days per week; OR
  * Beta agonist use on at least two days per week; OR
  * FEV1 < 85% predicted

Groups A & B:

Exclusion Criteria:

* Current smokers (smoking within the last 12 months) or former smokers who have a total pack-year smoking history greater than 10
* Pregnant women
* Subjects with a history of lung disease other than asthma
* Subjects with a history of a medical disease, which in the opinion of the investigator may put the subject at extra risk from study-related procedures or because the disease may influence the results of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prescott G Woodruff, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: UCSF Airway Clinical Research Center — http://acrc.ucsf.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Non-asthmatic Controls | Asthmatics (Treatment) | Asthmatics (no Treatment)
Started | 21 | 22 | 12
Completed | 20 | 19 | 10
Not Completed | 1 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The sample size for baseline analysis (n=50) does not match the overall enrolled participants (n=55) because the investigators only included samples for baseline analysis if participants completed all visits and had analyzable samples from those visits.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Non-asthmatic Controls | Asthmatics (Treatment) | Asthmatics (no Treatment) | Total
Number analyzed (Participants) | 20 | 19 | 11 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.05 (5.34) | 26.15 (5.01) | 32.72 (13.49) | 29.16 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 5 | 28
  Male | 9 | 7 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 1 | 8
  Not Hispanic or Latino | 15 | 12 | 8 | 35
  Unknown or Not Reported | 3 | 2 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 0 | 5
  White | 9 | 9 | 6 | 24
  More than one race | 0 | 3 | 0 | 3
  Unknown or Not Reported | 2 | 3 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 11 | 50
FEV1 [Mean (Standard Deviation); unit: liters] — The volume of air exhaled in the first second of a forced exhalation maneuver, in liters.
  liters | 3.68 (0.93) | 3.41 (1.01) | 3.52 (0.97) | 3.54 (0.99)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Baseline T Cell miRNA Expression Between Asthmatics and Healthy Controls
Description: Identification of T cell miRNAs which are differentially expressed in asthma as compared to healthy controls. The investigators will measure a panel of ~200 miRNAs by qPCR (yielding normalized copy numbers for each miR) and identify differential expressed based on a false discovery rate <0.05. Normalized copy numbers from this qPCR experiment were established using the "global mean-normalization" approach as described in the paper by Barbara D'haene et al. entitled "miRNA expression profiling - from reference genes to global mean normalization" published in MicroRNA Expression profiling Methods and Protocols, Springer Verlag, Feb 2011.
Time Frame: Baseline (cross-sectional analysis)
Population: The study enrolled two groups of subjects: 1. Healthy Non-asthmatic Controls, 2. Asthmatics (who were subsequently randomized to inhaled corticosteroids or no treatment). This analysis compares pre-randomization values in group 1 healthy non-asthmatics controls to group 2 asthmatics because the scientific goal is to identify miRNAs differentially expressed in asthma.
Measure: Mean (Standard Deviation); unit: Normalized log2 copy number
Groups:
- Healthy Non-asthmatic Controls: Healthy non-asthmatic controls who underwent bronchoscopy at one time point and served as a control group for the asthmatics group for evaluation of T-cell miRNA expression.
- Asthmatics (Baseline): All steroid-naïve asthmatics. These subjects were studied before and after randomization to study drug or no treatment. The pre-randomization data were collected on these asthmatics as one uniform group for comparison to healthy controls. These subjects then underwent bronchoscopy and T-cell miRNA measurement at pre-randomization and again 8 weeks after randomization to inhaled corticosteroids or no treatment.
Arm/Group | Healthy Non-asthmatic Controls | Asthmatics (Baseline)
Number analyzed (Participants) | 19 | 25
Normalized log2 copy number
  mir1: number analyzed (Participants) | 10 | 23
  mir1 | 13.2 (5.5) | 10.2 (3.0)
  mir107: number analyzed (Participants) | 12 | 21
  mir107 | 13.6 (4.5) | 11.7 (3.2)
  mir128: number analyzed (Participants) | 13 | 19
  mir128 | 17.0 (5.9) | 16.5 (3.9)
  mir141: number analyzed (Participants) | 12 | 19
  mir141 | 14.6 (4.5) | 13.3 (2.0)
  mir148b: number analyzed (Participants) | 17 | 22
  mir148b | 14.5 (5.2) | 11.9 (3.3)
  mir181b: number analyzed (Participants) | 15 | 19
  mir181b | 11.5 (5.5) | 10.8 (2.6)
  mir185: number analyzed (Participants) | 15 | 22
  mir185 | 12.7 (5.0) | 10.7 (2.4)
  mir194: number analyzed (Participants) | 10 | 21
  mir194 | 11.5 (8.1) | 8.7 (3.5)
  mir19a: number analyzed (Participants) | 10 | 20
  mir19a | 13.8 (7.1) | 10.4 (2.5)
  mir200a: number analyzed (Participants) | 11 | 19
  mir200a | 14.9 (7.2) | 14.9 (3.1)
  mir22: number analyzed (Participants) | 12 | 20
  mir22 | 14.2 (6.2) | 12.3 (2.9)
  mir223: number analyzed (Participants) | 10 | 20
  mir223 | 12.3 (4.6) | 10.7 (1.4)
  mir23a: number analyzed (Participants) | 8 | 20
  mir23a | 14.2 (5.0) | 13.6 (2.8)
  mir26a: number analyzed (Participants) | 7 | 20
  mir26a | 10.2 (6.7) | 9.4 (2.8)
  mir320b: number analyzed (Participants) | 14 | 19
  mir320b | 13.8 (3.4) | 12.4 (2.6)
  mir598: number analyzed (Participants) | 13 | 22
  mir598 | 12.4 (2.1) | 13.4 (2.2)
  mir720: number analyzed (Participants) | 14 | 23
  mir720 | 12.1 (5.2) | 11.6 (5.1)
  mir1915: number analyzed (Participants) | 14 | 23
  mir1915 | 7.7 (1.6) | 8.8 (1.1)
  mir1978: number analyzed (Participants) | 14 | 17
  mir1978 | 11.7 (3.7) | 13.1 (2.6)
Statistical Analysis 1: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir1; Test type: Superiority; p = 0.32, t-test, 2 sided — This p value is adjusted for multiple comparisons using the false discovery rate (FDR) approach and a p value <0.05 is taken for significance; Mean Difference (Net) = 3.04
Statistical Analysis 2: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir107; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.91
Statistical Analysis 3: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir128; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.47
Statistical Analysis 4: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir141; Test type: Superiority; p = 0.42, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.27
Statistical Analysis 5: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir148b; Test type: Superiority; p = 0.32, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.55
Statistical Analysis 6: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir181b; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.68
Statistical Analysis 7: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir185; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.94
Statistical Analysis 8: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir194; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.77
Statistical Analysis 9: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir19a; Test type: Superiority; p = 0.32, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.38
Statistical Analysis 10: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir200a; Test type: Superiority; p = 0.99, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.00
Statistical Analysis 11: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir22; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.92
Statistical Analysis 12: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir223; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.57
Statistical Analysis 13: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir23a; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.52
Statistical Analysis 14: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir26a; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.81
Statistical Analysis 15: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir320b; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.39
Statistical Analysis 16: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir598; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.92
Statistical Analysis 17: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir720; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.55
Statistical Analysis 18: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir1915; Test type: Superiority; p = 0.30, t-test, 2 sided; Mean Difference (Net) = -1.12
Statistical Analysis 19: Comparison: Healthy Non-asthmatic Controls vs Asthmatics (Baseline); mir1978; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.35

2. Primary Outcome: Change From Baseline of T Cell miRNA Expression at 8 Weeks in Asthmatics in Response to Inhaled Corticosteroids vs. no Treatment
Description: Identification of T cell miRNAs which were reduced in asthmatics who were randomized to inhaled corticosteroids as compared to those randomized to no treatment. The investigators will measure the same miRNAs by qPCR as identified in the other Primary Outcome and define a significant change using a multiple comparison adjusted p-value (false discovery rate <0.05).
Time Frame: 8 weeks after randomization to inhaled corticosteroids or no treatment
Population: This analysis population had two groups: 1. Asthmatics who were randomized to treatment with inhaled corticosteroids, 2. Asthmatics who were randomized to no treatment.
Measure: Mean (Standard Deviation); unit: Normalized log2 copy number
Groups:
- Asthmatics (Treatment): Asthmatics randomized to inhaled budesonide, 1 puff (180mcg) twice a day for 8-10 weeks. These subjects will undergo bronchoscopy and T-cell miRNA measurement at pre-randomization (before corticosteroids) and again after treatment with inhaled corticosteroids.
  Budesonide: Inhaled powder of inhaled corticosteroid, 1 puff (180mcg) twice a day for 8-10 weeks
- Asthmatics (no Treatment): Asthmatics randomized to no treatment with inhaled corticosteroids for 8-10 weeks. These subjects will undergo bronchoscopy and T-cell miRNA measurement at pre-randomization and again 8 weeks after randomization to no treatment with inhaled corticosteroids.
Arm/Group | Asthmatics (Treatment) | Asthmatics (no Treatment)
Number analyzed (Participants) | 14 | 7
Normalized log2 copy number
  mir1: number analyzed (Participants) | 13 | 7
  mir1 | 1.5 (4.6) | -3.0 (4.5)
  mir107: number analyzed (Participants) | 11 | 6
  mir107 | 0.86 (4.4) | -3.7 (4.0)
  mir128: number analyzed (Participants) | 10 | 5
  mir128 | 2.0 (3.6) | -1.6 (2.2)
  mir141: number analyzed (Participants) | 11 | 3
  mir141 | 1.2 (3.0) | 1.7 (3.7)
  mir148b: number analyzed (Participants) | 14 | 5
  mir148b | 1.5 (5.0) | -3.1 (4.4)
  mir181b: number analyzed (Participants) | 11 | 5
  mir181b | -0.12 (4.9) | -1.7 (4.3)
  mir185: number analyzed (Participants) | 10 | 6
  mir185 | 0.72 (3.8) | -2.2 (3.4)
  mir194: number analyzed (Participants) | 7 | 5
  mir194 | -0.73 (5.3) | -0.37 (2.8)
  mir19a: number analyzed (Participants) | 10 | 5
  mir19a | 0.053 (3.8) | -2.4 (3.0)
  mir200a: number analyzed (Participants) | 9 | 5
  mir200a | -1.4 (3.9) | -2.2 (2.4)
  mir22: number analyzed (Participants) | 8 | 5
  mir22 | 0.059 (4.6) | -2.7 (3.7)
  mir223: number analyzed (Participants) | 10 | 4
  mir223 | 0.90 (3.3) | -1.0 (3.0)
  mir23a: number analyzed (Participants) | 11 | 5
  mir23a | 1.5 (3.8) | -2.8 (1.5)
  mir26a: number analyzed (Participants) | 9 | 3
  mir26a | 1.2 (3.6) | -0.43 (5.4)
  mir320b: number analyzed (Participants) | 10 | 3
  mir320b | 0.86 (7.6) | 1.8 (3.7)
  mir598: number analyzed (Participants) | 14 | 5
  mir598 | -0.20 (3.3) | -3.5 (3.0)
  mir720: number analyzed (Participants) | 10 | 6
  mir720 | -1.9 (6.6) | -0.87 (4.3)
  mir1915: number analyzed (Participants) | 11 | 6
  mir1915 | -0.49 (2.1) | 0.26 (1.7)
  mir1978: number analyzed (Participants) | 10 | 5
  mir1978 | 2.3 (5.1) | -1.5 (2.5)
Statistical Analysis 1: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir1; Test type: Superiority; p = 0.26, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.53
Statistical Analysis 2: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir107; Test type: Superiority; p = 0.26, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.52
Statistical Analysis 3: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir128; Test type: Superiority; p = 0.26, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.57
Statistical Analysis 4: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir141; Test type: Superiority; p = 0.87, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.58
Statistical Analysis 5: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir148b; Test type: Superiority; p = 0.29, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.57
Statistical Analysis 6: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir181b; Test type: Superiority; p = 0.75, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.56
Statistical Analysis 7: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir185; Test type: Superiority; p = 0.36, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.90
Statistical Analysis 8: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir194; Test type: Superiority; p = 0.89, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.36
Statistical Analysis 9: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir19a; Test type: Superiority; p = 0.48, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.48
Statistical Analysis 10: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir200a; Test type: Superiority; p = 0.87, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.75
Statistical Analysis 11: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir22; Test type: Superiority; p = 0.53, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.78
Statistical Analysis 12: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir223; Test type: Superiority; p = 0.57, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.91
Statistical Analysis 13: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir23a; Test type: Superiority; p = 0.26, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.27
Statistical Analysis 14: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir26a; Test type: Superiority; p = 0.75, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.66
Statistical Analysis 15: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir320b; Test type: Superiority; p = 0.89, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.91
Statistical Analysis 16: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir598; Test type: Superiority; p = 0.26, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.32
Statistical Analysis 17: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir720; Test type: Superiority; p = 0.87, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.99
Statistical Analysis 18: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir1915; Test type: Superiority; p = 0.74, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.75
Statistical Analysis 19: Comparison: Asthmatics (Treatment) vs Asthmatics (no Treatment); mir1978; Test type: Superiority; p = 0.36, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.77

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events during their study participation, which ranged from 2 weeks to 10 weeks depending on the group to which they were assigned.
Arm/Group | Healthy Non-asthmatic Controls | Asthmatics (Treatment) | Asthmatics (no Treatment)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/22 | 0/12
Other Adverse Events (participants affected / at risk) | 3/21 | 1/22 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Non-asthmatic Controls (N=21) | Asthmatics (Treatment) (N=22) | Asthmatics (no Treatment) (N=12)
Medication error during bronchoscopy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — This event was unrelated to study drug. During a bronchoscopy, the participant was erroneously given epinephrine by the procedure nurse. This event was followed to completion and reported to the IRB, OHRP, sponsor, and medical center.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Non-asthmatic Controls (N=21) | Asthmatics (Treatment) (N=22) | Asthmatics (no Treatment) (N=12)
Decreased systolic blood pressure from sedation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Decreased lung function post-procedure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No